CLINICAL TRIAL: NCT00100620
Title: Efficacy and Safety of Zoledronic Acid in the Prevention and Treatment of Corticosteroid Induced Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446O2306
Record Dates: First submitted 2005-01-03; First posted 2005-01-04 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis
Keywords: Corticosteroid induced osteoporosis; prevention; treatment; zoledronic acid
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
The intake of high doses of corticosteroids is known to play an important role in the weakening of the bones and is thus an increasing fracture risk. Zoledronic acid (Aclasta) is a drug known for its protective effect in some bone diseases (tumors, paget). This study will test the safety and efficacy of zoledronic acid in the prevention and treatment of corticosteroid induced osteoporosis in male and female patients.

ELIGIBILITY:
Inclusion Criteria:

* Long duration treatment with corticosteroids (started or ongoing)

Exclusion Criteria:

* History of osteogenesis imperfecta, multiple myeloma or Paget's disease
* History of Hyperparathyroidism, hyperthyroidism
* History of Osteomalacia

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 802
Dates: Start 2004-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Percent change in lumbar spine Bone Mineral Density at Month 12 relative to baseline.

SECONDARY OUTCOMES:
Percent change in lumbar spine Bone Mineral Density at Month 6 relative to baseline
Percent change in total hip, femoral neck, trochanter and distal radius Bone Mineral Density at Months 6 and 12 relative to baseline
Biochemical markers of bone turnover at Baseline, Day 10, Month 3, Month 6, Month 12
Overal safety of zoledronic acid compared to risedronate in patients receiving corticosteroid therapy

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Center for Education and research on Therapeutics (CERTs) of Musculoskeletal Disorders, Birmingham, Alabama
  - United Osteoporosis Centers, Gainesville, Georgia
  - Osteoporosis & Clinical Trials, Cumberland, Maryland
  - University of Ohio, Columbus, Ohio
  - Radiant Research, Wyomissing, Pennsylvania
  - McGuire VA Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Devogelaer JP, Sambrook P, Reid DM, Goemaere S, Ish-Shalom S, Collette J, Su G, Bucci-Rechtweg C, Papanastasiou P, Reginster JY. Effect on bone turnover markers of once-yearly intravenous infusion of zoledronic acid versus daily oral risedronate in patients treated with glucocorticoids. Rheumatology (Oxford). 2013 Jun;52(6):1058-69. doi: 10.1093/rheumatology/kes410. Epub 2013 Jan 30. PMID 23365149
- [Derived] Grbic JT, Black DM, Lyles KW, Reid DM, Orwoll E, McClung M, Bucci-Rechtweg C, Su G. The incidence of osteonecrosis of the jaw in patients receiving 5 milligrams of zoledronic acid: data from the health outcomes and reduced incidence with zoledronic acid once yearly clinical trials program. J Am Dent Assoc. 2010 Nov;141(11):1365-70. doi: 10.14219/jada.archive.2010.0082. PMID 21037195
- [Derived] Reid DM, Devogelaer JP, Saag K, Roux C, Lau CS, Reginster JY, Papanastasiou P, Ferreira A, Hartl F, Fashola T, Mesenbrink P, Sambrook PN; HORIZON investigators. Zoledronic acid and risedronate in the prevention and treatment of glucocorticoid-induced osteoporosis (HORIZON): a multicentre, double-blind, double-dummy, randomised controlled trial. Lancet. 2009 Apr 11;373(9671):1253-63. doi: 10.1016/S0140-6736(09)60250-6. PMID 19362675